CLINICAL TRIAL: NCT02513303
Title: A Phase 3, Randomized, Multicenter, Single-blind, Controlled Study Evaluating Arteriovenous Fistula Outcomes With and Without a Perivascular Sirolimus-Eluting Collagen Implant
Brief Title: Trial to Evaluate the Sirolimus-Eluting Collagen Implant on AV Fistula Outcomes
Acronym: ACCESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vascular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VT-304
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Complication of Renal Dialysis; End Stage Renal Disease; End Stage Kidney Disease; ESRD; Chronic Kidney Failure; Complication of Hemodialysis; Vascular Access Complication; Arteriovenous Fistula
Keywords: Dialysis; End Stage Renal Disease; End Stage Kidney Disease; ESRD; Chronic Kidney Failure; Chronic Renal Failure; Chronic Kidney Disease; Hemodialysis; Vascular Access; Arteriovenous Fistula; AV Fistula; AVF; Nephrology; Vascular Surgery; Dialysis Access
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula; Renal Insufficiency, Chronic | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): AV fistula surgery Single administration of sirolimus-eluting Collagen implant
  Interventions: Drug: Sirolimus; Procedure: AV Fistula Surgery; Device: Sirolimus-eluting Collagen Implant (SeCI)
- Control Group (Other): AV fistula surgery
  Interventions: Procedure: AV Fistula Surgery

INTERVENTIONS:
Drug: Sirolimus — A single dose of sirolimus delivered locally
  Other Names: Rapamycin
  Arms: Treatment Group
Procedure: AV Fistula Surgery — AV Fistula Surgery
Device: Sirolimus-eluting Collagen Implant (SeCI) — SeCI placed at and around the site of the anastomosis of an AV fistula, immediately following completion of a successful AV fistula surgery.
  Other Names: Rapamycin
  Arms: Treatment Group

SUMMARY:
The objective of this study is to evaluate efficacy and safety outcomes following use of the Sirolimus-eluting Collagen Implant (SeCI) in subjects undergoing surgical creation of an AV fistula for vascular access (index procedure).

DETAILED DESCRIPTION:
The objective of this study is to evaluate efficacy and safety outcomes following use of the Sirolimus-eluting Collagen Implant (SeCI) in subjects undergoing surgical creation of an AV fistula for vascular access (index procedure). Following successful creation of the AV fistula, the cohort randomized to the treatment group will receive the SeCI; the control group will not receive an implant. The primary hypothesis is that the proportion of subjects that meet requirements for fistula suitability for dialysis six months following the index procedure will be higher in the treatment group in comparison to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Currently on hemodialysis for ≤12 months or expected to initiate hemodialysis within approximately 6 months of the creation of the AV fistula.
* Vascular anatomy suitable for creation of the AV fistula, determined by pre procedure duplex ultrasound
* Successful creation of a single stage radiocephalic or brachiocephalic end to side fistula

Exclusion Criteria:

* Prior AV access created on the limb where the fistula surgery is planned
* ST-elevation MI or cerebrovascular accident within 30 days of the index procedure
* Known hypersensitivity to the following: sirolimus, beef or bovine collagen
* Hypotension with systolic blood pressures <100 mm Hg at the time of screening
* Known or suspected active infection at the time of the AV fistula surgery
* Known to be HIV positive
* Prisoner, mentally incompetent, and/or alcohol or drug abuser

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2015-11; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Iyer, MD, Study Director — Vascular Therapies, Inc.
Locations (4):
- United States (4):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - AKDHC Medical Research Service, Phoenix, Arizona
  - San Diego Institute of Medical Research, Escondido, California
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirogen: Participants received single administration of Sirolimus-eluting Collagen Implant (Sirogen) at the time of AV fistula surgery
- Control: Participants underwent AV fistula surgery without an implant
- Run-in: Participants received single administration of Sirolimus-eluting Collagen Implant (Sirogen) at the time of AV fistula surgery. The first subject enrolled by a participating surgeon was a run-in subject; run-in subjects were part of the randomized set; all run-in subjects receive Sirogen.
Period: Overall Study
Arm/Group | Sirogen | Control | Run-in
Started | 125 | 118 | 26
Completed | 105 | 101 | 22
Not Completed | 20 | 17 | 4
Not completed — Withdrawal by Subject | 9 | 7 | 2
Not completed — Lost to Follow-up | 2 | 4 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Death | 8 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirogen | Control | Run-in | Total
Number analyzed (Participants) | 125 | 118 | 26 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 74 | 82 | 13 | 169
  >=65 years | 51 | 36 | 13 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (14.9) | 57.7 (13.9) | 61.4 (17.3) | 59.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 6 | 57
  Male | 97 | 95 | 20 | 212
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 8 | 3 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 31 | 30 | 8 | 69
  White | 84 | 81 | 15 | 180
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 125 | 118 | 26 | 269
Kidney Disease Status at Enrollment [Count of Participants; unit: Participants]
  Chronic kidney disease | 33 | 36 | 1 | 70
  End stage renal disease | 92 | 82 | 25 | 199

OUTCOME MEASURES:

1. Primary Outcome: Fistula Suitability for Dialysis at 6 Months (FSD6)
Description: For subjects who are on hemodialysis by day 150, suitability for dialysis will be determined by the ability to use the fistula for dialysis using 2-needles with a mean dialysis machine blood pump speed of ≥300 mL/min for two-thirds of the dialysis sessions during a 30 day suitability ascertainment period that begins 150 days after fistula creation.
  For subjects who are not on hemodialysis on day of enrollment and who do not initiate hemodialysis by day 150, suitability for dialysis will be determined by a vascular ultrasound performed at the 6 month follow up visit. Suitability for dialysis will be defined as a fistula with an access vein diameter (AVD) of ≥6 mm (internal diameter) and an access blood flow of ≥500 mL/min.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirogen | Control | Run-in
Number analyzed (Participants) | 125 | 118 | 26
Participants
  Met FSD6 criteria | 74 | 76 | 21
  Did not meet FSD6 criteria | 43 | 35 | 5
  Indeterminant FSD6 | 8 | 7 | 0
Statistical Analysis 1: Comparison: Sirogen vs Control; Test type: Superiority; p = 0.2942, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 1 year
Description: The safety set for adverse event reporting comprises of patients assigned to control arm having received investigational product.
Arm/Group | Sirogen | Control | Run-in
All-Cause Mortality (participants affected / at risk) | 8/127 | 4/116 | 2/26
Serious Adverse Events (participants affected / at risk) | 56/127 | 55/116 | 15/26
Other Adverse Events (participants affected / at risk) | 115/127 | 101/116 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirogen (N=127) | Control (N=116) | Run-in (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0 | 2
Cardiac failure acute (Cardiac disorders) | 1 | 5 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 7 | 3 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 1 | 0
Coronary ostial stenosis (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 1
Chest pain (General disorders) | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 1 | 0
Cystitis bacterial (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 1
Pleural infection bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 6 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 3
Septic shock (Infections and infestations) | 2 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 2 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4 | 3 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 3 | 5 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 6 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 3
Uraemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 3 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
End stage renal disease (Renal and urinary disorders) | 2 | 5 | 3
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Refusal of treatment by patient (Social circumstances) | 2 | 0 | 0
Atrial septal defect repair (Surgical and medical procedures) | 0 | 1 | 0
Renal transplant (Surgical and medical procedures) | 2 | 2 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypertensive crisis (Vascular disorders) | 2 | 4 | 1
Hypertensive emergency (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Steal syndrome (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirogen (N=127) | Control (N=116) | Run-in (N=26)
Vision blurred (Eye disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 1
Nausea (Gastrointestinal disorders) | 9 | 4 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 3 | 7 | 4
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 71 | 59 | 14
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 17 | 18 | 6
Haemodialysis complication (Injury, poisoning and procedural complications) | 41 | 35 | 6
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 11 | 6 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 8 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 6 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Dizziness (Nervous system disorders) | 7 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Hypotension (Vascular disorders) | 3 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT02513303/Prot_SAP_000.pdf